CLINICAL TRIAL: NCT03649763
Title: Onset and Duration of Forearm Nerve Blockade Performed With a Single Distal Injection Versus Sequential Injections at Distal and Proximal Locations Alongside the Nerves: A Blinded Randomized
Brief Title: Onset and Duration of Forearm Nerve Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York School of Regional Anesthesia (Other)
Responsible Party: Principal Investigator, Catherine Vandepitte, M.D., Medical Doctor, New York School of Regional Anesthesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1801
Record Dates: First submitted 2018-08-01; First posted 2018-08-28 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lidocaine distal forearm (Active Comparator): Lidocaine 1% - Ultrasound-guided specific blocks of the DISTAL median and ulnar nerves with perineural injections of Lidocaine1%. Volume injected is 6 mL/nerve; 12 mL total.
  Interventions: Drug: Lidocaine
- Bupivacaine distal forearm (Active Comparator): Bupivacaine 0.5%-Ultrasound-guided specific blocks of the DISTAL median and ulnar nerves with perineural injections of Bupivacaine0.5%. Volume injected is 6 mL/nerve; 12 mL total.
  Interventions: Drug: Bupivacaine
- Lidocaine distal and proximal forearm (Active Comparator): Lidocaine 1%- Ultrasound-guided specific blocks of the DISTAL and PROXIMAL median and ulnar nerves with perineural injections of Lidocaine 1%. Volume injected is 3 mL/nerve; 12 mL total
  Interventions: Drug: Lidocaine
- Bupivacaine distal and proximal forearm (Active Comparator): Bupivacaine 0.5%- Ultrasound-guided specific blocks of the DISTAL and PROXIMAL median and ulnar nerves with perineural injections of Bupivacaine 0.5 %. Volume injected is 3 mL/nerve; 12 mL total.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Lidocaine — lidocaine 1%, distal ( ulnar and medial nerve): 6ml/nerve , 12m total
  Arms: Lidocaine distal forearm
Drug: Bupivacaine — Bupivacaine 0.5%,distal ( ulnar and medial nerve): 6ml/nerve , 12m total
  Arms: Bupivacaine distal and proximal forearm; Bupivacaine distal forearm
Drug: Lidocaine — lidocaine 1%, distal and proximal ( ulnar and medial nerve): 3ml/nerve , 12m total
  Arms: Lidocaine distal and proximal forearm

SUMMARY:
This pilot study will evaluate the latency of onset and duration of sensory-motor block in patients undergoing hand surgery. Patients will be randomized to receive nerve blocks of the distal forearm or of the distal and proximal forearm. Local anesthetic will be injected to anesthetise the median and ulnar nerves in the distal forearm (1-injection site group) or the median and ulnar nerves in the distal and proximal forearm (2-sequential injection sites group) to accomplish anesthesia for surgery on the hand.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo daycare surgery for carpal tunnel syndrome under peripheral nerve blocks
* American Society of Anesthesiologists (ASA) physical status I, II or III
* Able to demonstrate sensory function in the ulnar and median nerve distribution by exhibiting sensitivity to cold, pinprick and light touch
* Scheduled to undergo primary hand surgery
* Able to understand the Dutch language, purpose and risks of the study
* Able to provide informed consent and authorization to use protected health information, adhere to the study visit schedule, and complete all study assessments

Exclusion Criteria:

* Currently pregnant or nursing
* History of hypersensitivity to local anesthetics
* Contraindication to lidocaine, bupivacaine, paracetamol
* Medical condition that will make it difficult to assess sensory distributions of the upper extremity peripheral nerves or to communicate with staff
* Suspected or known recent history (< 3 months) of drug or alcohol abuse
* Concurrent physical condition that may require analgesic treatment (such as NSAID or opioid) in the postsurgical period for pain that is not strictly related to Carpal Tunnel Syndrome and which may confound the postsurgical assessments
* Infection at the planned block site(s)
* Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®)
* Body weight <40 kg or body mass index >44 kg/m2
* Uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments
* Any chronic neuromuscular deficit affecting the Ulnar and Median nerves or muscles of the surgical extremity
* Any chronic condition or disease that would compromise neurological
* Presence of pre-existing coagulation disorders
* Baseline neurological deficits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 5-minute beginning at the end of the last injection
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 10-minute beginning at the end of the last injection
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 15-minute beginning at the end of the last injection
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 20-minute beginning at the end of the last injection
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 25-minute beginning at the end of the last injection
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 30-minute beginning at the end of the last injection
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 45-minute beginning at the end of the last injection
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 60-minute beginning at the end of the last injection
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | Post Anesthesia Care Unit arrival
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 15-minute after Post Anesthesia Care Unit arrival
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | 30-minute after Post Anesthesia Care Unit arrival
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.
onset of successful block and duration of sensory-motor blockade of the median and ulnar nerves | Post Anesthesia Care Unit discharge
  Block success is defined as full sensory block of the areas and muscles supplied by the median and ulnar nerves. Block failure is defined as absence of sensory blockade at 30 min in the median and ulnar nerve territories as assessed by pin-prick, cold and light touch.

SECONDARY OUTCOMES:
postoperative Numeric Rating Scale (NRS) | screening Day0 (prior to the nerve block), post block, PACU arrival, Day0 evening, Day1 morning and evening, Day2 morning and evening, Day3 morning and evening, Day4, Day5, Day6, Day7
  pain rating(numeric rating scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | post block
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Post Anesthesia Care Unit arrival
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 0 evening
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 1 morning
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 1 evening
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 2 morning
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 2 evening
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 3 morning
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 3 evening
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 4
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 5
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 6
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 7
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)
postoperative Numeric Rating Scale (NRS) | Day 30
  pain rating( Numeric Rating Scale) at rest and with movement ( scale 0:no pain - 10:worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided